CLINICAL TRIAL: NCT04452500
Title: Phase IIa Trial of a Selective Glucocorticoid Receptor Antagonist in the Treatment of Veterans With Posttraumatic Stress Disorder (PTSD)
Brief Title: Phase IIa Trial of a Selective Glucocorticoid Receptor Antagonist in the Treatment of Veterans With Posttraumatic Stress Disorder (PTSD) (Seven Study)
Acronym: SEVEN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHBB-014-18S; CX001917-01 (Other Grant/Funding Number: VA CSR&D)
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: PTSD
Keywords: Glucocorticoids; Posttraumatic Stress Disorder; Quality of Life
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — CORT 108297

STUDY DESIGN:
Intervention Model Description: The investigators propose a two-site parallel group, randomized, double-blind, placebo-controlled Phase IIa clinical trial to test the efficacy and safety of CORT108297- 180mg daily for 7 days for PTSD symptoms in Veterans.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CORT108297 (Experimental): CORT108297- 180mg daily for 7 days
  Interventions: Drug: CORT108297
- Placebo (Placebo Comparator): Placebo- 180mg daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CORT108297 — CORT108297- 180mg daily for 7 days
  Arms: CORT108297
Drug: Placebo — Placebo- 180mg daily for 7 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the drug CORT108297, which blocks the hormone cortisol, for treatment of PTSD in Veterans, and establish a safety profile that will inform the design of future studies.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase IIa clinical trial to test the efficacy and safety of CORT108297- 180mg daily for 7 days for PTSD symptoms in Veterans. Each of the two sites will enroll 44 Veterans with chronic PTSD. Participants first will undergo screening procedures, including a clinical psychological interview, self-report questionnaires, blood draw, and medical evaluations. If eligible, they will be randomized to either CORT108297 or placebo. The same procedures will be repeated at several in-person and virtual visits before, during and after taking the study drug or placebo for seven days. The key outcome measures will be obtained at baseline, day 7, 28, and day 56.

There is large body of evidence demonstrating that Posttraumatic Stress Disorder (PTSD) is associated with alterations in the stress hormone cortisol. There is also evidence that medications that block cortisol may be beneficial for treating PTSD and depression. This study will test a medication, CORT108297, which is from a new class of cortisol blockers which have no effect on other hormones. CORT108297 has been shown to have efficacy in preclinical CNS models and was well tolerated and safe in Phase I healthy volunteer studies making it a candidate for further development. Thus, the goal will be to complete a Phase IIa proof of concept trial of CORT108297 to focus on safety and tolerability and obtain pilot efficacy data to inform the design of future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* History of US military service
* Capable of reading and understanding English
* Able to provide written informed consent
* Symptoms of PTSD (must score 23 or greater on the CAPS-5 assessment at screening visit)
* Men and pre-menopausal women must agree to use two forms of reliable contraception, one of which is a barrier method.
* Participants who use an SSRI or SNRI medication for PTSD must be on a stable dose for 8 weeks before enrollment.
* Participants who use trazodone for sleep must be on a stable dose.
* Participants who use opiate pain medication must be on a stable dose.
* For participants who are in psychotherapy, treatment must be stable for 6 weeks.

Exclusion Criteria:

* Alcohol use that meets criteria for Alcohol Use Disorder in past 3 months.
* Marijuana or other drug use that meets criteria for Substance Use Disorder in past 3 months.
* Ever diagnosed with: Bipolar Disorder, Schizophrenia, Schizoaffective Disorder, Obsessive-Compulsive Disorder, or Major Depressive Disorder with Psychotic Features
* Experienced any psychologically traumatic event in the past 3 months
* Currently using certain antidepressant medications such as doxepin or tricyclics
* Currently using certain mood stabilizers, such as lithium
* Currently using antipsychotic medication
* High risk for suicide or violent behavior
* Has sleep apnea and not using any treatment, such as CPAP
* Currently using corticosteroid medication (oral or inhaled)
* History of neurological disease
* Angina, congestive heart failure or low blood pressure
* Heart attack in the past 6 months
* Heart block or irregular heartbeat
* Kidney failure, liver failure or pancreatitis
* Severe chronic obstructive pulmonary disease (COPD)
* History of liver disease with lab results on AST or ALT more than 2 times the normal readings
* History of kidney disease with lab results on eGFR less than 60 ml/min
* History of additional risk factors for Torsades de pointes, such as heart failure, low potassium, or family history of a heart rhythm disorder called long QT syndrome
* Use of certain medications that can affect heart rhythm
* Use of certain medications that can interfere with the effects of the study drug
* High blood pressure that is not controlled by medication
* Diabetes that is not well-controlled
* History of certain types of head injuries
* Mild cognitive impairment

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 (CAPS) | 56 days
  The CAPS is a 30-item interview that is the gold standard assessment for PTSD. The CAPS provides a dimensional and categorical measure of PTSD, and incorporates frequency and intensity of symptoms into a single severity score.
Frequency, Intensity, Burden of Side Effects (FIBSER) | 56 days
  The FIBSER is a self-report 0-6 Likert-type scale that measures global frequency, intensity, and overall burden of side effects.

SECONDARY OUTCOMES:
Columbia Suicide Severity Rating Scale | 56 days
  The C-SSRS is FDA approved for assessing severity and change of suicidality in drug studies.
PTSD Checklist for DSM-5 | 56 days
  The PCL is a validated self-report scale assessing PTSD symptoms corresponding to DSM-5.
World Health Organization Quality of Life (WHOQOL-BREF) | 56 days
  The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original WHOQOL-100 instrument and is more convenient for use in large research studies or clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Neylan, MD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (2):
- United States (2):
  - Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
For the proposed work final de-identified data from this project will be shared as widely as possible with the scientific community using UCSF DataShare (aka Dash). This self-service tool, available to any UCSF affiliated researcher, is a collaboration between University of California San Francisco's Library, and the UC Curation Center (UC3) at the California Digital Library and the UCSF Clinical and Translational Science Institute (CTSI).
Supporting Information: SAP, CSR
Time Frame: Within 1 year of the end of the funding period.
Access Criteria: After the raw data is made available on the Dash site, anyone will also be able to view the descriptive metadata used to index the data set. This information is publicly available to allow for maximum discoverability. Individuals wishing to access the data must agree to terms of use for the data set via a Data Use Agreement, and may have to meet additional requirements as set forth by the PI. The data will be permanently archived and available through the California Digital Library.